CLINICAL TRIAL: NCT00660062
Title: Relapse Prevention in Patients With a Major Depressive Episode Treated With Electroconvulsive Treatment Using a Fixed Dose Range of Escitalopram Compared to a Fixed Dose of Nortriptyline (DUAG-7) A Randomised Controlled 6 Month Double-blind Study
Brief Title: Relapse Prevention With Escitalopram or Nortriptyline Following Electro-Convulsive Treatment (DUAG-7)
Acronym: DUAG-7
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow inclusion
Sponsor: Hillerod Hospital, Denmark (Other)
Responsible Party: Principal Investigator, Klaus Martiny, Senior Consultant, Hillerod Hospital, Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DUAG-7
Record Dates: First submitted 2008-04-14; First posted 2008-04-17 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2011-04

CONDITIONS: Major Depression
Keywords: Major depression; relapse prevention; ECT; escitalopram; nortriptyline
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram; Nortriptyline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Escitalopram 10 mg daily (Experimental): Escitalopram 10 mg daily
  Interventions: Drug: escitalopram
- Escitalopram 20 mg daily (Experimental): Escitalopram 20 mg daily
  Interventions: Drug: escitalopram
- escitalopram 30 mg daily (Experimental): escitalopram 30 mg daily
  Interventions: Drug: escitalopram
- Nortriptylin 100 mg daily (Active Comparator): Nortriptylin 100 mg daily
  Interventions: Drug: nortriptyline

INTERVENTIONS:
Drug: escitalopram — 10 mg daily
  Arms: Escitalopram 10 mg daily
Drug: escitalopram — 20 mg daily dosage
  Arms: Escitalopram 20 mg daily
Drug: escitalopram — 30 mg daily dosage
  Arms: escitalopram 30 mg daily
Drug: nortriptyline — 100 mg daily dosage
  Arms: Nortriptylin 100 mg daily

SUMMARY:
The main purpose of this study is to investigate the relapse preventing efficacy of escitalopram in a dose range and nortriptylin in a single dose in patients having been treated successfully with a course of electroconvulsive treatment (ECT).

DETAILED DESCRIPTION:
This study records severity of depression and relapse in patients treated for a major depressive disorder with electroconvulsive treatment (ECT)in a period og 6 month after end of ECT treatment. Patients will be randomized into four groups treated with escitalopram 10 mg, 20 mg, 30 mg or nortriptylin 100 mg daily dosages. The primary outcome measure is relapse and secondary outcome measure is tolerability.

The study is a multicenter trial within Denmark.

ELIGIBILITY:
Inclusion Criteria:

* Remission from a major depressive episode after ECT treatment

Exclusion Criteria:

* Suicidality (Hamilton item 3 score of 3 or more)
* Symptoms mania (MAS score of 15 or more)
* Duration of actual depressive episode more than 2 years
* Compulsory measures of any kind
* Dementia
* Severe somatic illness
* Pregnant or lactating subject
* Known clinical relevant malabsorption.
* Epilepsia
* Clinically substantial cognitive deterioration due to ECT treatment
* schizophrenia, schizopreniform or schizo-affective disorder
* Bipolar I, Bipolar II eller
* Rapid cycling bipolar disorder
* Abuse of alcohol or drugs
* Early relapse (less than 2 month) after ECT
* Inadequate contraception
* Known intolerance to any of the used study medications
* Myocardial infarction in the last 6 month
* Clinical important liver disease
* Any known disturbance of the cardiac conduction system, cardiac insufficiency,or other clinical important cardiac disease
* Treatment with a MAO-inhibitor
* Treatment with norepinephrine or epinephrine
* Known hyperthyroidism or treatment with thyroid hormones
* Known ortostatic hypertension.
* Glaucoma
* Known hereditary galactoseintolerance, Lapp Lactase deficiency) or gluco-se/galactosemalabsorption.
* Ongoing treatment with sympatomimetica efedrine, isoprenaline, physostigmine, dopamine, levodopa, phenylephrine.
* Ongoing treatment with anticholinergica, antiparkinson treatment, antihistamines, atropine, biperiden,
* Ongoing treatment with drugs that prolongs the cardiac QT-interval, such as quinidine, antihistamines, terfenadine og sotalole
* Ongoing treatment with fluconazole or terbinafine
* Ongoing treatment with mefloquin.
* Known intolerance to escitalopram
* Ongoing treatment with serotonergic acting substances such as tramadole, sumatriptane

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2009-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Hamilton depression rating scale | 14 days

SECONDARY OUTCOMES:
Drop out due to side-effects of drugs | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Martiny, MD,PhD, Principal Investigator — Mental Health Center Copenhagen Department O
Locations (1):
- Mental Health Centre Copenhagen Department O, Copenhagenl, Denmark

REFERENCES:
- [Background] Sackeim HA, Haskett RF, Mulsant BH, Thase ME, Mann JJ, Pettinati HM, Greenberg RM, Crowe RR, Cooper TB, Prudic J. Continuation pharmacotherapy in the prevention of relapse following electroconvulsive therapy: a randomized controlled trial. JAMA. 2001 Mar 14;285(10):1299-307. doi: 10.1001/jama.285.10.1299. PMID 11255384
- [Derived] Martiny K, Larsen ER, Licht RW, Nielsen CT, Damkier P, Refsgaard E, Lunde M, Straaso B, Christensen EM, Lolk A, Holmskov J, Sorensen CH, Brodsgaard I, Eftekhari SZ, Bendsen BB, Klysner R, Terp IM, Larsen JK, Vestergaard P, Buchholtz PE, Gram LF, Bech P; Danish University Antidepressant Group (DUAG*). Relapse Prevention in Major Depressive Disorder After Successful Acute Electroconvulsive Treatment: a 6-month Double-blind Comparison of Three Fixed Dosages of Escitalopram and a Fixed Dose of Nortriptyline - Lessons from a Failed Randomised Trial of the Danish University Antidepressant Group (DUAG-7). Pharmacopsychiatry. 2015 Nov;48(7):274-8. doi: 10.1055/s-0035-1565063. Epub 2015 Nov 3. PMID 26529118